CLINICAL TRIAL: NCT00209222
Title: Efficacy of 6x R-CHOP Followed by Myeloablative Radiochemotherapy and Autologous Stem Cell Transplantation vs. 3 x (R-CHOP/R-DHAP) Followed by a High Dose ARA-C Containing Myeloablative Regimen and Autologous Stem Cell Transplantation
Brief Title: Efficacy of R-CHOP vs R-CHOP/R-DHAP in Untreated MCL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Mantle Cell Lymphoma Network (Other)
Collaborators: German Low Grade Lymphoma Study Group (Other); Lymphoma Study Association (Other)
Responsible Party: Prof Dr. Martin Dreyling, University Hospital Grosshadern/European MCLNetwork
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCL2004-2
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2009-07

CONDITIONS: Lymphoma, Mantle-Cell
Keywords: Lymphoma, Mantle-Cell; younger patients; chemotherapy; high dose therapy; C04.557.386.480.300.725.500; C15.604.515.569.480.300.725.500; C20.683.515.761.480.300.725.500
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Cisplatin; Cytarabine; Dexamethasone; Carmustine; Melphalan; Etoposide; Granulocyte Colony-Stimulating Factor; R-CHOP protocol; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): induction: R-CHOP consoldiation : TBI/Cyclo
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: BCNU; Drug: Melphalan; Drug: Etoposide; Drug: G-CSF; Procedure: chemotherapy: R-CHOP; Procedure: chemotherapy: Dexa-BEAM; Procedure: stem cell harvest; Procedure: total body irradiation; Procedure: high-dose chemotherapy: Cyclophosphamide
- 2 (Experimental): induction: R-CHOP/DHAP consolditaion: TBI/TAM
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Cisplatinum; Drug: Ara-C; Drug: Dexamethasone; Drug: Melphalan; Drug: G-CSF; Procedure: chemotherapy: R-CHOP; Procedure: chemotherapy: R-DHAP; Procedure: stem cell harvest; Procedure: total body irradiation; Procedure: high-dose chemotherapy: Ara-C /Melphalan

INTERVENTIONS:
Drug: Rituximab — antibody
Drug: Cyclophosphamide — chemotherapy
Drug: Doxorubicin — chemotherapy
Drug: Vincristine — chemotherapy
Drug: Prednisone — corticosteroide
Drug: Cisplatinum — chemotherapy
  Arms: 2
Drug: Ara-C — chemotherapy
  Arms: 2
Drug: Dexamethasone — corticosteroide
  Arms: 2
Drug: BCNU — chemotherapy
  Arms: 1
Drug: Melphalan — chemotherapy
Drug: Etoposide — chemotherapy
  Arms: 1
Drug: G-CSF — growth factor
Procedure: chemotherapy: R-CHOP — immuno-chemotherapy
Procedure: chemotherapy: R-DHAP — immuno-chemotherapy
  Arms: 2
Procedure: chemotherapy: Dexa-BEAM — chemotherapy
  Arms: 1
Procedure: stem cell harvest — procedure
Procedure: total body irradiation — radiation
Procedure: high-dose chemotherapy: Cyclophosphamide — chemotherapy
  Arms: 1
Procedure: high-dose chemotherapy: Ara-C /Melphalan — chemotherapy
  Arms: 2

SUMMARY:
The aim of this study is to determine whether alternating courses of cyclophosphamide, doxorubicin, vincristine, prednisone/dexamethasone, cytarabine, cisplatin (CHOP/DHAP) plus rituximab followed by total body irradiation [TBI]/high dose cytarabine [ARA-C]/melphalan-peripheral blood stem cell transplantation (TAM-PBSCT) can improve the time to treatment failure compared to CHOP plus rituximab followed by standard PBSCT (dexamethasone, carmustine, cytarabine, etoposide, and melphalan [Dexa-BEAM]/TBI/high dose cyclophosphamide) in patients with untreated mantle cell lymphoma.

DETAILED DESCRIPTION:
Recently, a prospective randomized intergroup trial of the European MCL Network has shown that a myeloablative radio-chemotherapy followed by autologous stem cell transplantation (PBSCT) improves event-free survival (EFS) when compared to a interferon alpha maintenance therapy after a CHOP-like induction. However, the CR rate after the CHOP induction was still low (<20%). Thus, several studies have been conducted to increase the CR rate of induction therapy to further improve event-free and overall survival. Two recent phase II trials suggest that induction regimens containing high dose Ara-C may significantly improve the CR rate up to 80%. In addition, a number of studies provide evidence that the humanized anti-CD20 antibody Rituximab may induce significant responses in relapsed MCL. A prospective randomized study of the GLSG demonstrated that a combined immuno-chemotherapy (CHOP plus Rituximab) induces a significantly higher response rate than CHOP alone.

The aim of this study is the comparison of the current standard (R-CHOP followed by myeloablative radio-chemotherapy and subsequent blood stem cell transplantation) to a new alternating induction regimen containing high dose Ara-C (R-CHOP/DHAP) followed by a high dose ARA-C containing myeloablative radio-chemotherapy and PBSCT.

This study will be performed as a prospective, randomized, open-label multicenter phase III trial. All patients will be initial randomized for standard treatment versus experimental treatment.

REFERENCE ARM:

The induction therapy consists of 6 cycles of a CHOP chemotherapy in combination with Rituximab. If the mantle cell lymphoma is progressive after 4 cycles of chemotherapy, patients will be taken off study. Patients achieving at least a partial remission after 6 cycles R-CHOP will proceed to intensified consolidation (Dexa-BEAM) with stem cell collection and subsequent myelo-ablative radio-chemotherapy (TBI/High Dose Cyclophosphamide) with autologous stem cells transplantation

EXPERIMENTAL ARM:

Initial cytoreductive chemotherapy comprises of alternating cycles of 3xCHOP and 3x DHAP plus Rituximab. Patients with progressive disease after 2 treatment cycles R-CHOP and 2x R-DHAP will be off study. Patients achieving at least a partial remission after 3x CHOP and 3x DHAP plus Rituximab will proceed to with stem cell collection. The subsequent myeloablative radio-chemotherapy with stem cell transplantation consists of a radiotherapy (TBI), high dose Ara-C and Melphalan.

The primary end point in this study is the time to treatment failure. The time to treatment failure will be defined as time from start of initial therapy until first failure. A failure will be defined as failure of initial therapy or progression of the lymphoma or death of the patient.

Using the data of the PBSCT group in the former European mantle cell study as baseline in a proportional hazard model, the improvement for the time to treatment failure expected by the new strategy can be expressed by reduction of relative risk (rr). A risk reduction to 52% which would correspond to a improvement of 20% in failure free survival after 3 years seems to be a clinical relevant improvement. For a working significance level alpha=0.05 and a power of 95% the number of events necessary for a one sided fixed sample trial is about 105. During this study the time to treatment failure will be monitored using an equivalent one-sided triangular sequential test.

In order to evaluate the impact of therapy on overall survival in this patients, a total follow up of about 12 years for this study is expected.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of mantle cell lymphoma (World Health Organization [WHO] classification)
* Clinical stage II - IV (Ann Arbor)
* Previously untreated patients
* Age 18 - 65 years
* WHO performance < 2
* Measurable disease (also: patients with isolated bone marrow involvement)
* Informed consent according to International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use/European Union Good Clinical Practice (ICH/EU GCP) and national/local regulations

Exclusion Criteria:

* Age > 65 years
* WHO performance status > 2
* Known anti-murine antibody (HAMA) reactivity or known hypersensitivity to murine antibodies
* Previous lymphoma therapy with radiation, cytostatic drugs, anti-CD20 antibody or interferon
* Serious disease interfering with a regular therapy according to the study protocol:

  * cardiac (e.g. manifest heart failure, coronary heart disease, uncontrolled hypertension)
  * pulmonary (e.g. chronic lung disease with hypoxemia)
  * endocrine (e.g. severe, not sufficiently controlled diabetes mellitus)
  * renal insufficiency (unless caused by the lymphoma): creatinine > 2x normal value and/or creatinine clearance < 50 ml/min)
  * impairment of liver function (unless caused by the lymphoma): transaminases > 3x normal or bilirubin > 2,0 mg/dl
* Patients with unresolved hepatitis B or C infection or known HIV infection
* Prior organ, bone marrow or peripheral blood stem cell transplantation
* Concomitant or previous malignancies within the last 5 years other than basal cell skin cancer or in situ uterine cervix cancer.
* Pregnancy or lactation
* Any psychological, familiar, sociological, or geographical condition potentially hampering compliance with the study protocol and follow up schedule

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2004-07; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
time to treatment failure after start of therapy

SECONDARY OUTCOMES:
complete remission (CR) rate
overall survival
progression-free survival
adverse events
serious infectious complications

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hermine, PhD, Principal Investigator — University Hospital Necker, Dept. of Adult Hematology; Wolfgang Hiddemann, PhD, Study Chair — University Hospital Großhadern/LMU, Dept. of Medicine III
Locations (3):
- Groupe D´Etudes des Lymphomes De l´Adulte (GELA), Paris, France
- German Low Grade Study Group (Glsg), Munich, Germany
- The Maria Sklodowska Memorial, Cancer Center - Inst. of Oncology, Warsaw, Poland

REFERENCES:
- [Background] Dreyling M, Lenz G, Hoster E, Van Hoof A, Gisselbrecht C, Schmits R, Metzner B, Truemper L, Reiser M, Steinhauer H, Boiron JM, Boogaerts MA, Aldaoud A, Silingardi V, Kluin-Nelemans HC, Hasford J, Parwaresch R, Unterhalt M, Hiddemann W. Early consolidation by myeloablative radiochemotherapy followed by autologous stem cell transplantation in first remission significantly prolongs progression-free survival in mantle-cell lymphoma: results of a prospective randomized trial of the European MCL Network. Blood. 2005 Apr 1;105(7):2677-84. doi: 10.1182/blood-2004-10-3883. Epub 2004 Dec 9. PMID 15591112
- [Background] Lenz G, Dreyling M, Hoster E, Wormann B, Duhrsen U, Metzner B, Eimermacher H, Neubauer A, Wandt H, Steinhauer H, Martin S, Heidemann E, Aldaoud A, Parwaresch R, Hasford J, Unterhalt M, Hiddemann W. Immunochemotherapy with rituximab and cyclophosphamide, doxorubicin, vincristine, and prednisone significantly improves response and time to treatment failure, but not long-term outcome in patients with previously untreated mantle cell lymphoma: results of a prospective randomized trial of the German Low Grade Lymphoma Study Group (GLSG). J Clin Oncol. 2005 Mar 20;23(9):1984-92. doi: 10.1200/JCO.2005.08.133. Epub 2005 Jan 24. PMID 15668467
- [Derived] Hermine O, Jiang L, Walewski J, Bosly A, Thieblemont C, Szymczyk M, Pott C, Salles G, Feugier P, Hubel K, Haioun C, Casasnovas RO, Schmidt C, Bouabdallah K, Ribrag V, Kanz L, Durig J, Metzner B, Sibon D, Cheminant M, Burroni B, Klapper W, Hiddemann W, Unterhalt M, Hoster E, Dreyling M; European Mantle Cell Lymphoma Network. High-Dose Cytarabine and Autologous Stem-Cell Transplantation in Mantle Cell Lymphoma: Long-Term Follow-Up of the Randomized Mantle Cell Lymphoma Younger Trial of the European Mantle Cell Lymphoma Network. J Clin Oncol. 2023 Jan 20;41(3):479-484. doi: 10.1200/JCO.22.01780. Epub 2022 Dec 5. PMID 36469833
- [Derived] Hermine O, Hoster E, Walewski J, Bosly A, Stilgenbauer S, Thieblemont C, Szymczyk M, Bouabdallah R, Kneba M, Hallek M, Salles G, Feugier P, Ribrag V, Birkmann J, Forstpointner R, Haioun C, Hanel M, Casasnovas RO, Finke J, Peter N, Bouabdallah K, Sebban C, Fischer T, Duhrsen U, Metzner B, Maschmeyer G, Kanz L, Schmidt C, Delarue R, Brousse N, Klapper W, Macintyre E, Delfau-Larue MH, Pott C, Hiddemann W, Unterhalt M, Dreyling M; European Mantle Cell Lymphoma Network. Addition of high-dose cytarabine to immunochemotherapy before autologous stem-cell transplantation in patients aged 65 years or younger with mantle cell lymphoma (MCL Younger): a randomised, open-label, phase 3 trial of the European Mantle Cell Lymphoma Network. Lancet. 2016 Aug 6;388(10044):565-75. doi: 10.1016/S0140-6736(16)00739-X. Epub 2016 Jun 14. PMID 27313086
- [Derived] Delfau-Larue MH, Klapper W, Berger F, Jardin F, Briere J, Salles G, Casasnovas O, Feugier P, Haioun C, Ribrag V, Thieblemont C, Unterhalt M, Dreyling M, Macintyre E, Pott C, Hermine O, Hoster E; European Mantle Cell Lymphoma Network. High-dose cytarabine does not overcome the adverse prognostic value of CDKN2A and TP53 deletions in mantle cell lymphoma. Blood. 2015 Jul 30;126(5):604-11. doi: 10.1182/blood-2015-02-628792. Epub 2015 May 28. PMID 26022239
- [Derived] Hoster E, Klapper W, Hermine O, Kluin-Nelemans HC, Walewski J, van Hoof A, Trneny M, Geisler CH, Di Raimondo F, Szymczyk M, Stilgenbauer S, Thieblemont C, Hallek M, Forstpointner R, Pott C, Ribrag V, Doorduijn J, Hiddemann W, Dreyling MH, Unterhalt M. Confirmation of the mantle-cell lymphoma International Prognostic Index in randomized trials of the European Mantle-Cell Lymphoma Network. J Clin Oncol. 2014 May 1;32(13):1338-46. doi: 10.1200/JCO.2013.52.2466. Epub 2014 Mar 31. PMID 24687837
- [Derived] Pott C, Hoster E, Delfau-Larue MH, Beldjord K, Bottcher S, Asnafi V, Plonquet A, Siebert R, Callet-Bauchu E, Andersen N, van Dongen JJ, Klapper W, Berger F, Ribrag V, van Hoof AL, Trneny M, Walewski J, Dreger P, Unterhalt M, Hiddemann W, Kneba M, Kluin-Nelemans HC, Hermine O, Macintyre E, Dreyling M. Molecular remission is an independent predictor of clinical outcome in patients with mantle cell lymphoma after combined immunochemotherapy: a European MCL intergroup study. Blood. 2010 Apr 22;115(16):3215-23. doi: 10.1182/blood-2009-06-230250. Epub 2009 Dec 23. PMID 20032498